CLINICAL TRIAL: NCT03586180
Title: Medical Clowning: Needs Assessment, Implication, and Evaluation for Children and Adolescents With Cancer Using Child Friendly Healthcare
Brief Title: Medical Clowning: Needs Assessment and Implication for Hospitalized Children With Cancer/Blood Disease
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201803121RINB
Record Dates: First submitted 2018-06-04; First posted 2018-07-13 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-05

CONDITIONS: Blood Disease; Cancer; Friendly Healthcare in Children; Medical Clown; Hospitalized Children
MeSH Terms: conditions — Hematologic Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children and their parents: aged 4-18 children with cancer/blood disease and their parents
  Interventions: Behavioral: Medical Clowning for children
- Dr. Clowns: they will perform shows for children and parents
  Interventions: Behavioral: Medical Clowning for children

INTERVENTIONS:
Behavioral: Medical Clowning for children — Clowns in clinical setting have been found to be effective in reducing children's experiences of these effects during hospitalization and before procedures.

SUMMARY:
Hospitalized children who undergo painful procedures are more susceptible than others to experiencing iatrogenic effects, such as anxiety, pain, and severe stress. Clowns in clinical setting have been found to be effective in reducing children's experiences of these effects during hospitalization and before procedures. This article provides an overview of clowning in health care settings; reviews major studies conducted on clowning for hospitalized children, discussing evidence that clown interventions decrease pain and distress in pediatric patients; and concludes with a discussion of health care clowning as a profession.

ELIGIBILITY:
Inclusion Criteria:

* aged 4-18 children with cancer/blood disease and parents of children aged 0-18 years with cancer/blood disease

Exclusion Criteria:

* older than aged 18

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: aged 4-18 children with cancer/blood disease and parents of children aged 0-18 years with cancer/blood disease
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
experience and influence from medical clowning for children and their parents | 1 year
  Children with cancer/blood disease and their parents would use self-report to complete the questionnaire after medical clowning. Using Face Rating Scale (1=very unhappy to 5=very happy) for measuring emotion state (pre-emotion for before medical clowning and post-emotion for after medical clowning). It can understand whether their emotion state change before/after medical clowning or not.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Universtiy Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided